CLINICAL TRIAL: NCT00797680
Title: Duration of Hypothermia for Neuroprotection After Pediatric Cardiac Arrest
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Laerdal Medical (Industry)
Responsible Party: Principal Investigator, Ericka Fink, Associate Professor, Pediatric Critical Care Medicine, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ef1; K23NS065132 (NIH)
Record Dates: First submitted 2008-11-24; First posted 2008-11-25 (Estimated); Last update posted 2016-01-18 (Estimated); Status verified 2016-01

CONDITIONS: Cardiac Arrest; Brain Injury
Keywords: Pediatric cardiac arrest
MeSH Terms: conditions — Heart Arrest; Brain Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 72 hours hypothermia (Experimental): 72 hours hypothermia
  Interventions: Other: 72 hours hypothermia
- 24 hours hypothermia (Experimental): 24 hours hypothermia
  Interventions: Other: 24 hours hypothermia

INTERVENTIONS:
Other: 72 hours hypothermia — 72 hours mild hypothermia (33 +/1 1 degree Celsius)
  Arms: 72 hours hypothermia
Other: 24 hours hypothermia — 24 hours mild hypothermia (33 +/1 1 degree Celsius)
  Arms: 24 hours hypothermia

SUMMARY:
In this study, children who survive cardiac arrest will be evaluated whether 24 or 72 hours of whole body hypothermia (cooling) during recovery is better to help prevent brain injury and improve outcome. The investigators will also test the safety of cooling patients for 24 and 72 hours. The investigators hypothesize that 72 hours of cooling will be more beneficial than 24 hours without compromising safety.

DETAILED DESCRIPTION:
Cooling has been shown to decrease the amount of brain injury that can occur after heart attacks in adults and in newborn babies with birth asphyxia (a lack of blood flow and oxygen to the fetus). It is unknown if cooling is effective in children after cardiac arrest. However, cooling is recommended by the American Heart Association as a "consideration" for use in children after cardiac arrest to prevent brain injury and has been used by doctors in our intensive care unit since 2002.

Children will be randomly assigned to receive either 24 or 72 hours of cooling and compare the results of 1) blood-and urine derived markers of brain injury, and 2) brain magnetic resonance imaging and spectroscopy (MRI and MRS), which measures the anatomy and chemical patterns in the brain without using ionizing radiation, between the two groups of patients with 24 or 72 hours of cooling. We will also evaluate if cooling has any effect on patient outcome and quality of life at 6 months and one year using telephone or mail questionnaires.

A child may take part in this research study if he or she had a cardiac arrest, received help with breathing and chest compressions to get a spontaneous heart rate by a health care worker, and remains unconscious in the intensive care unit (ICU). The attending physician in the ICU has already decided to cool your child to provide protection for his or her brain function.

Children invited to participate in this study also are between 1 week and 17 years of age, have access tubes already in place in an artery or vein for blood draws, a urine catheter, are able to undergo MRI and MRS brain scans, and, if female, cannot be pregnant.

Patients can not have had an acute brain injury from other causes (ex., meningitis, trauma), hemorrhage (excess bleeding from any site), congenital heart disease, do not resuscitate status, are undergoing a brain death examination, or have a known coagulation defect that makes them bleed more easily. The study will be performed on a total of 40 children strictly in this hospital.

ELIGIBILITY:
Inclusion Criteria:

* Chest compressions by a health care worker Age 1 wk - 17 yr ROSC attained PICU attending decides to cool Central venous or arterial catheter Glasgow Coma Score ≤ 8

Exclusion Criteria:

Other acute brain injury (TBI, meningitis) Do not resuscitate status Pregnancy Absolute contraindication to MRI Brain death evaluation Metabolic disorder Active hemorrhage Pre-existing coagulation defect

Ages: 1 Week to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2008-10; Primary Completion 2014-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Degree of brain injury as measured by serum and urine biomarkers and Magnetic Resonance Spectroscopy | hospital discharge

SECONDARY OUTCOMES:
Frequency of adverse events | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Ericka L Fink, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Kernan KF, Berger RP, Clark RSB, Scott Watson R, Angus DC, Panigrahy A, Callaway CW, Bell MJ, Kochanek PM, Fink EL, Simon DW. An exploratory assessment of serum biomarkers of post-cardiac arrest syndrome in children. Resuscitation. 2021 Oct;167:307-316. doi: 10.1016/j.resuscitation.2021.07.007. Epub 2021 Jul 14. PMID 34271122
- [Derived] Fink EL, Wisnowski J, Clark R, Berger RP, Fabio A, Furtado A, Narayan S, Angus DC, Watson RS, Wang C, Callaway CW, Bell MJ, Kochanek PM, Bluml S, Panigrahy A. Brain MR imaging and spectroscopy for outcome prognostication after pediatric cardiac arrest. Resuscitation. 2020 Dec;157:185-194. doi: 10.1016/j.resuscitation.2020.06.033. Epub 2020 Jul 9. PMID 32653571